CLINICAL TRIAL: NCT02541487
Title: Fetal Effects of Pre-Pregnancy Lifestyle Interventions in Unexplained Infertility Patients
Status: Completed | Type: Observational
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Other Study IDs: Fit-Later
Record Dates: First submitted 2015-08-18; First posted 2015-09-04 (Estimated); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A de-identified sample of blood will be collected at the time of the baseline visit.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Nutritional/Physical Activity (NuPA) Intervention: Obese participants in the FIT-PLESE clinical trial randomized to the nutritional restriction /AlliTM/physical activity arm that achieve pregnancy.
  Interventions: Dietary Supplement: Alli-nutritional supplement
- Physical Activity only (PAo) Intervention: Obese participants in the FIT-PLESE clinical trial randomized to the exercise only arm that achieve pregnancy.
- Infertile, non-lifestyle intervention controls: Obese women (60) with unexplained infertility who meet the inclusion/exclusion criteria for FIT-PLESE but decline participation in the trial and who elect to undergo CC-IUI treatment and achieve pregnancy without prior diet and exercise interventions.

INTERVENTIONS:
Dietary Supplement: Alli-nutritional supplement — Obese participants in the FIT-PLESE clinical trial randomized to the nutritional restriction /AlliTM/physical activity arm that achieve pregnancy.
  Groups: Nutritional/Physical Activity (NuPA) Intervention

SUMMARY:
This is a cross-sectional comparison study of three maternal and fetal groups. Patients studied are women (and their fetus if they conceive) participating in the Reproductive Medicine Network's (RMN) FIT-PLESE investigation (funded, the NuPA and PAo arms) compared to control mothers who decline the intervention protocols and their fetuses if they conceive.

DETAILED DESCRIPTION:
Via participation in the FIT-PLESE study (from the RMN) we will randomize 90 obese women with unexplained infertility 1:1 to a lifestyle modification program consisting of nutritionally balanced caloric restriction (1200-1500 kcal/d), a gastric lipase inhibitor (Alli) and increased physical activity (with a goal of reaching 10K steps/d) (NuPA) versus increased physical activity alone (PAo). The pre-pregnancy intervention lasts 16 weeks, with a goal of 7% weight loss in the NuPA arm. Weight and physical activity are monitored with wireless devices (Fitbit Wireless Activity Tracker and Fitbit Aria Wireless Activity Scale, respectively). Following the 16 week pre-pregnancy intervention, all randomized couples will undergo standard treatment for unexplained infertility, 3 cycles of CC-IUI (requiring ~3 months). The goal for both treatment groups is to maintain levels of physical activity and weight achieved during the pretreatment phase during the empiric infertility treatment phase. Women who conceive will be followed throughout pregnancy with the wireless activity monitors and wireless scales. Additionally there will be three brief onsite visits during pregnancy (at 16, 24 and 32 weeks) for determination of weight, waist circumference, glycemic measures (fasting glucose, insulin, and HgbA1C), apolipoprotein lipids, and blood pressure. Nutritional intake will be assessed with The Dietary Assessment Questionnaire and Diet History Questionnaire II (DHQ II), the instrument chosen by FIT-PLESE investigators (http://appliedresearch.cancer.gov/dhq2/). The primary outcomes of FIT-PLESE are the live-birth rate, birth weight, gestational age at delivery, and congenital anomaly rate. The subject inclusion and exclusion criteria are detailed in the Human Subjects section. There is no overlap between the aims of FIT-PLESE and those of the present R21 proposal.

The three maternal and fetal groups for this proposal are as follows:

FIT-PLESE participants (University of Pennsylvania Central IRB approved)

Group 1: Nutritional/Physical Activity (NuPA) Intervention: Obese participants in the FIT-PLESE clinical trial randomized to the nutritional restriction /AlliTM/physical activity arm that achieve pregnancy.

Group 2: Physical Activity only (PAo) Intervention: Obese participants in the FIT-PLESE clinical trial randomized to the exercise only arm that achieve pregnancy.

Control group (University of Oklahoma IRB approved) Group 3 (Infertile, non-lifestyle intervention controls): Obese women (60) with unexplained infertility who meet the inclusion/exclusion criteria for FIT-PLESE but decline participation in the trial and who elect to undergo CC-IUI treatment and achieve pregnancy without prior diet and exercise interventions.

We have extensive experience evaluating fetal morphometry from women participating in a prospective study designed to assess the relationship between maternal and neonatal adiposity (n=77) who have already undergone similar ultrasound and biomarker measurements during pregnancy at OUHSC. The data have been collected and are being analyzed. These non-diabetic women with uncomplicated pregnancies were evenly distributed between pre-pregnancy BMIs for normal weight (BMI <24.9, n=23), overweight (BMI 25-29.9, n=29) or obese (BMI 30>, n=25). These women conceived spontaneously and did not undergo diet or exercise intervention (see preliminary data below).

We will assess participants of Group 1, 2 and 3 prior to pregnancy and during each trimester at 16, 24, and 32 weeks gestational age for the mothers who conceive. We will then evaluate each fetus of those who conceive during each trimester of pregnancy at the same gestational ages. We will evaluate newborns within one week of delivery for body composition. All participants will have the same inclusion and exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 18 to ≤ 40 years of age, with one or more years infertility history, desirous of conceiving, regularly ovulating (defined as 9 or more menses per year), at initiation of participation.
* BMI ≥ 30 kg/m2 obtained at screening visit.
* Normal uterine cavity and at least one open fallopian tube confirmed by hysterosalpingography (HSG), sonohysterography (SHG), or laparoscopy/hysteroscopy in the last three years preceding enrollment into the study. An uncomplicated intrauterine non-IVF pregnancy and uncomplicated delivery and postpartum course resulting in live birth within the last three years will also serve as sufficient evidence of a patent tube and normal uterine cavity as long as the subject did not have, during the pregnancy or subsequently, risk factors for Asherman's syndrome or tubal disease or other disorder leading to an increased suspicion for intrauterine abnormality or tubal occlusion.
* Evidence of ovarian function/reserve as assessed by day 3 (+/-2 days) FSH ≤ 10 IU/L with Estradiol ≤ 70 pg/mL OR AMH ≥ 1 ng/mL within one year prior to study initiation.
* Normal or corrected thyroid function within one year of study initiation.
* Normal or corrected prolactin level within one year of study initiation.
* In general good health, not taking any medications which could interfere with the study (e.g., FSH, insulin sensitizers).
* Ability to have inseminations following hCG administration
* Male partner with total motile sperm in the ejaculate of at least 5 million sperm, within one year of study initiation
* Able to comply with intercourse instructions and collection of semen for insemination
* Anyone enrolled and randomized to the RMN FIT PLESE study

Exclusion Criteria:

* Currently pregnant or successful pregnancies within 12 months of initiating participation. Clinical intrauterine miscarriages prior to initiating participation, within ASRM guidelines: subjects over 35 must wait six months, while subjects under 35 must wait 12 months. No exclusion for biochemical pregnancies.
* Undiagnosed abnormal uterine bleeding.
* Suspicious ovarian mass.
* Subjects on oral contraceptives, depo-progestins, or hormonal implants (including Implanon). A two month washout period will be required prior to screening for patients on these agents. Longer washouts may be necessary for certain depot contraceptive forms or implants, especially when the implants are still in place. A one-month washout will be required for patients who have taken oral cyclic progestins.
* Known 21-hydroxylase deficiency or other enzyme defect causing congenital adrenal hyperplasia.
* Type I or Type II diabetes mellitus, or if receiving antidiabetic medications.
* Known significant anemia (Hemoglobin <10 g/dL).
* History of deep venous thrombosis, pulmonary embolus, or cerebrovascular event.
* Known heart disease (New York Heart Association Class II or higher).
* Known liver disease (defined as AST or ALT >2 times normal, or total bilirubin >2.5 mg/dL).
* Known renal disease (defined as BUN >30 mg/dL or serum creatinine > 1.4 mg/dL).
* History of, or suspected cervical carcinoma, endometrial carcinoma or breast carcinoma.
* History of alcohol abuse (defined as >14 drinks/week) or binge drinking of ≥ 6 drinks at one time).
* Known Cushing's disease.
* Known or suspected adrenal or ovarian androgen secreting tumors.
* Allergy, known hypersensitivity or contraindication to the treatment medications used in this study including clomiphene citrate (previous change in vision).
* Couples with previous sterilization procedures (e.g. vasectomy, tubal ligation) whether or not it has been reversed.
* Subjects with untreated poorly controlled hypertension defined as a systolic blood pressure ≥ 160 mm Hg or a diastolic ≥ 100 mm Hg obtained on two measures obtained at least 60 minutes apart.
* Subjects who have undergone a bariatric surgery procedure in the past or are in a period of acute weight loss (defined as a weight loss of greater than 5 kgs in the last 6 months).
* Known moderate or severe endometriosis
* Anovulation or oligo-ovulation including hypothalamic amenorrhea, polycystic ovary syndrome, etc.
* Donated semen.
* Couples in which either partner is legally married to someone else.
* Medical conditions that are contraindications to pregnancy.
* Presence of severe, untreated psychiatric illness (major depression, substance abuse, eating disorder, etc.) that would, in the opinion of the site investigator, interfere with the patient's ability to successfully complete the study.
* Currently participating in a lifestyle intervention program (such as Weight Watchers, Atkins Diet, Curves) or lost more than 5% body weight within the last 6 months.
* History of Gout.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women that are seen in the OU Reproductive Medicine clinic.
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2015-05-08 (Actual); Primary Completion 2020-08-25 (Actual); Study Completion 2020-08-25 (Actual)

PRIMARY OUTCOMES:
evaluate fetal biometry | during pregnancy
evaluate subcutaneous abdominal, thigh, and arm adiposity. | during pregnancy
Placental volume will be determined | during pregnancy
Newborn body composition will be assessed with air displacement plethysmography (Pea Pod ®). | one week post-birth

CONTACTS AND LOCATIONS:
Overall Officials: Karl Hansen, MD, Principal Investigator — University of Oklahoma